CLINICAL TRIAL: NCT07249346
Title: An Open Label, Non-Randomized, Multi-Center Pilot Dose-Expansion Study of Low Dose Post-Transplant Cyclophosphamide/Tacrolimus/Ruxolitinib for GVHD Prophylaxis in Myeloablative Allogeneic Peripheral Blood Stem Cell Transplantation
Brief Title: Dose-Expansion Study of Low Dose Post-Transplant Cyclophosphamide/Tacrolimus/Ruxolitinib for Graft-versus-Host Disease (GVHD) Prophylaxis in Myeloablative Allogeneic Peripheral Blood Stem Cell Transplantation
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hannah Choe, MD (Other)
Collaborators: Incyte Corporation (Industry)
Responsible Party: Sponsor-Investigator, Hannah Choe, MD, Principal Investigator, Ohio State University Comprehensive Cancer Center
Organization: Ohio State University Comprehensive Cancer Center (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: OSU-24102
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Leukemia; Myelodysplasia; Chronic Myelomonocytic Leukemia
MeSH Terms: conditions — Leukemia; Anemia, Refractory, with Excess of Blasts; Leukemia, Myelomonocytic, Chronic | interventions — ruxolitinib; Hematopoietic Stem Cell Transplantation; Cyclophosphamide; Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Feasibility) (Experimental): Patients will receive post-transplant cyclophosphamide 25 mg/kg on Days +3 and +4, tacrolimus, and ruxolitinib for GVHD prophylaxis. Ruxolitinib will be dosed as ruxolitinib IR 5 mg po qD (on fluconazole, 5 mg po BID not on fluconazole) starting Day -1 until Day +28 and neutrophil engraftment and then increase to ruxolitinib IR 5 mg po BID (on fluconazole,10 mg po BID not on fluconazole) for up to 12 months. Tacrolimus will be tapered after Day +90 per institutional guidelines.
  Patients will receive ruxolitinib up to Day 180 posttransplant. Ruxolitinib will be tapered over 2-3 months depending on the starting dose at time of taper.
  Interventions: Drug: Ruxolitinib; Drug: Myeloablative conditioning regimen; Procedure: Hematopoietic Stem Cell Transplantation; Drug: Cyclophosphamide; Drug: Tacrolimus
- Cohort 2 (dose expansion) (Experimental): Patients will receive post-transplant cyclophosphamide 25 mg/kg on Days +3 and +4, tacrolimus, and ruxolitinib for GVHD prophylaxis. Ruxolitinib will be dosed as ruxolitinib IR 5 mg po qD (on fluconazole, 5 mg po BID not on fluconazole) starting Day -1 until Day +28 and neutrophil engraftment and then increase to ruxolitinib IR 5 mg po BID (on fluconazole,10 mg po BID not on fluconazole) for up to 12 months. Tacrolimus will be tapered after Day +90 per institutional guidelines.
  Patients will receive ruxolitinib up to Day 365 post-transplant. Ruxolitinib will be tapered over 2-3 months depending on the starting dose at time of taper.
  Interventions: Drug: Ruxolitinib; Drug: Myeloablative conditioning regimen; Procedure: Hematopoietic Stem Cell Transplantation; Drug: Cyclophosphamide; Drug: Tacrolimus

INTERVENTIONS:
Drug: Ruxolitinib — Taken PO
Drug: Myeloablative conditioning regimen — Patients will receive a full-intensity myeloablative conditioning regimen. Allowed regimens include:
  * Flu/Bu(130 mg/m2/day x 4 days)
  * Flu/TBI (8-12Gy)
  * Flu/Bu/Thiotepa The addition of alemtuzumab or ATG is not allowed.
Procedure: Hematopoietic Stem Cell Transplantation — Patients will undergo HCT
  Other Names: HCT
Drug: Cyclophosphamide — Given IV
Drug: Tacrolimus — Given PO

SUMMARY:
This is an open label, non-randomized, multicenter, pilot, dose expansion study of low dose post-transplant cyclophosphamide (25 mg/kg on Days +3 and +4)/tacrolimus/ruxolitinib in the setting of myeloablative conditioning (MAC) allogeneic peripheral blood stem cell transplantation (PBSCT).

DETAILED DESCRIPTION:
Primary Objective:

To assess survival without severe Grade 3-4 acute GVHD at Day 180 post-transplant in patients treated with GVHD prophylaxis in myeloablative allogeneic hematopoietic stem cell transplantation for patients treated with low dose PTCy(Cyclophosphamide)/Tac(Tacrolimus)/Rux(Ruxolitinib).

Secondary Objectives:

To describe rates of Grade II-IV and Grades III-IV acute GVHD, chronic GVHD requiring immunosuppression, hematologic recovery (neutrophil and platelet), disease relapse or progression, rates of Grade 3+ toxicity, primary and secondary graft failure, and overall survival (OS) for patients treated with low dose PTCy/Tac/Rux.

ELIGIBILITY:
Inclusion Criteria:

* Age 18.0 years or older at the time of enrollment
* Patients undergoing allogeneic hematopoietic cell transplantation for one of the following indications:

  * Acute leukemia with no circulating blasts and with less than 5% blasts in the bone marrow
  * Myelodysplasia/chronic myelomonocytic leukemia with no circulating blasts and with less than 10% blasts in the bone marrow (higher blast percentage allowed in MDS due to lack of differences in outcomes with <5% versus 5-10% blasts in this disease).

    * Planned myeloablative (MAC) conditioning regimen (see eligible regimens in Section 9.2)
* Patients must have a related or unrelated peripheral blood stem cell donor as follows:

  * Sibling donor must be a 6/6 match for HLA-A and -B at intermediate (or higher) resolution, and -DRB1 at high resolution using DNA-based typing and must be willing to donate peripheral blood stem cells and meet institutional criteria for donation.
  * Unrelated donor must be an 8/8 match at HLA-A, -B, -C and -DRB1 at high resolution using DNA-based typing.

Unrelated donor must be willing to donate peripheral blood stem cells and meet National Marrow Donor Program (NMDP) criteria for donation.

* Donor selection must comply with 21 CFR 1271

* Cardiac function: Left ventricular ejection fraction at least 45%
* Estimated creatinine clearance greater than 60 ml/min (C-G formula)
* Pulmonary function: DLCO (diffusing capacity of lung for carbon monoxide) corrected for hemoglobin at least 60% and FEV1 (forced expiratory volume at one second) predicted at least 60%
* Liver function: AST(Aspartate aminotransferase)/ALT(Alanine aminotransferase) <3x Upper Limit of Normal (ULN); Total bilirubin <2 mg/dL excluding Gilbert's syndrome or hemolysis
* Karnofsky Performance Score at least 70%.
* Female patients (unless postmenopausal for at least 1 year before the screening visit, or surgically sterilized), agree to practice two (2) effective methods of contraception at the same time, or agree to completely abstain from heterosexual intercourse, from the time of signing the informed consent through 12 months post-transplant.
* Male patients (even if surgically sterilized), of partners of women of childbearing potential must agree to one of the following: practice effective barrier contraception or abstain from heterosexual intercourse from the time of signing the informed consent through 12 months post-transplant.
* Plans for the use of targeted small molecule inhibitor post-transplant maintenance therapy must be disclosed upon enrollment. Planned use of investigational maintenance agents is not permitted. Planned hypomethylating agents as maintenance therapy is not permitted.

Allowed maintenance includes:

* FLT3 inhibitors: gilteritinib, sorafenib, midostaurin
* IDH inhibitors: enasidenib, ivosidenib
* BCR/ABL inhibitors: imatinib, ponatinib, dasatinib, nilotinib

  * Other targeted therapies may be discussed with protocol chairsVoluntary written consent obtained prior to the performance of any study-related procedure that is not a part of standard medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to future medical care.
  * There are no restrictions based on blood counts as this intervention is being used in combination with intensive chemotherapy with intent to myeloablate.

Exclusion Criteria:

* Prior allogeneic transplant
* Active CNS (central nervous system) involvement by malignant cells
* Patients with secondary acute myeloid leukemia arising from myeloproliferative neoplasms or overlap syndromes, including CMML(chronic myelomonocytic leukemia) and MDS/MPN (myelodysplastic syndromes/myeloproliferative neoplasms) syndromes; patients with secondary acute myeloid leukemia arising from myelodysplastic neoplasm are eligible.
* Patients with uncontrolled bacterial, viral, or fungal infections (currently taking medication and with progression or no clinical improvement) at time of enrollment.
* Active or inadequately treated latent infection with Mycobacterium tuberculosis (i.e., TB).
* Patients seropositive for human immunodeficiency virus (HIV) with detectable viral load. HIV+ patients with an undetectable viral load on antiviral therapy are eligible.
* Evidence of uncontrolled hepatitis B virus (HBV) or hepatitis C virus (HCV). The study allows:

  * Positive HBV serology with undetectable viral load and ongoing antiviral prophylaxis to prevent potential HBV reactivation.
  * Positive HCV serology with quantitative PCR (polymerase chain reaction) for plasma HCV RNA below the lower limit of detection, with or without concurrent antiviral HCV treatment.
* Arterial or venous thrombosis including DVT (deep vein thrombois), PE (pulmonary embolism), stroke, and myocardial infarction within six (6) months prior to enrollment or New York Heart Association (NYHA) Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia. Catheter-associated DVT is not exclusionary.
* Female patients who are pregnant or lactating
* Patients with a serious medical or psychiatric illness likely to interfere with participation in this clinical study
* Patients with prior malignancies except resected non-melanoma skin cancer or treated cervical carcinoma in situ. Cancer treated with curative intent ≥ 5 years previously will be allowed. Cancer treated with curative intent < 5 years previously must be reviewed and approved by the Protocol Officer or Chairs, qualifying as below.

  * the participant has been disease-free for at least 2 years and is deemed by the investigator to be at low risk of recurrence of that malignancy, or
  * the cancer has been deemed indolent with no progression over the last 2 years, and deemed by the investigator to be at low risk for further progression during the course of study and follow-up
  * the only prior malignancy was cervical cancer in situ and/or basal cell or squamous cell carcinoma of the skin
* Planned use of ATG or alemtuzumab in conditioning regimen
* Planned use of prophylactic donor leukocyte infusions
* Prior use of ruxolitinib
* Prior use of immune checkpoint inhibitors (i.e., PD1, PDL1, CTLA4 modulators) within six (6) months prior to conditioning
* History of congenital Long QT syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2026-06-01 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Severe acute GVHD-free Survival (SGFS) | At day 180 post-transplant
  SGFS will be calculated from the time of transplant to onset of grade 3-4 acute GVHD or death censoring patients alive without grade 3-4 GVHD at last clinical assessment date. The SGFS rate together with 95% confidence interval at day 180 will be estimated by Kaplan-Meier method.

SECONDARY OUTCOMES:
GVHD, relapse free survival (GRFS) | At 6 months and 1 year
  GVHD-free, relapse-free survival as a time to event outcome is defined as Grade III-IV acute GVHD, chronic GVHD requiring systemic immune suppression, underlying disease relapse or progression, or death by any cause.
Grade II-IV acute GVHD and Grade III-IV acute GVHD | At 6 months
  Cumulative incidences of Grade II-IV and III-IV acute GVHD will be determined. Acute GVHD will be graded according to standard MAGIC criteria. The time of onset of acute Grades II-IV and III-IV acute GVHD will be recorded, as well as the maximum grade achieved. Within the participants experiencing Grade II-IV acute GVHD, the proportion of patients with visceral involvement (liver or gut) will be described. Cumulative incidences of Minnesota standard and high risk acute GVHD will also be determined.
Chronic GVHD requiring immunosuppression | At 1 year
  Rate of chronic GVHD requiring immunosupression at 1 year
GVHD Free Survival (GFS) | At 1 year
  Events for this time to event outcome is defined as any of the following: 1) Grade III-IV acute GVHD, 2) chronic GVHD requiring systemic immune suppression, or 3) death by any cause. The time to the event is defined as the time to the earliest of the qualifying events. Subjects alive without experiencing an event will be censored at last available GVHD assessment
Hematologic Recovery (Neutrophil Counts) | Up to 2 years post transplant
  Hematologic recovery will be assessed according to neutrophil and platelet counts recovery after transplant. Neutrophil recovery is defined as achieving an absolute neutrophil count (ANC) greater than or equal to 500/mm3 for three consecutive measurements on three different days. The first of the three days will be designated the day of neutrophil recovery. The competing event is death or subsequent transplant without neutrophil recovery. For patients who never drop ANC below 500/mm3, the date of neutrophil recovery will be Day +1 post-transplant.
Disease Relapse or Progression | At 1 year
  Number of patients with disease relapse or progression. Relapse is defined by either morphological or cytogenetic evidence of acute leukemia or MDS consistent with pre-transplant features.
  Relapse will be diagnosed when there is:
  * Reappearance of leukemia blast cells in the peripheral blood; or,
  * Greater than 5% blasts in the bone marrow, not attributable to another cause (e.g., bone marrow regeneration); or, Page 56 of 63
  * The appearance of previous or new dysplastic changes (MDS specific) within the bone marrow with falling donor chimerism; or,
  * The development of extramedullary leukemia or leukemic cells in the cerebral spinal fluid or,
  * The reappearance of cytogenetic abnormalities present prior to transplantation
Non-relapse Mortality (NRM) | At 1 year
  The cumulative incidence of NRM will be estimated after hematopoietic cell transplantation (HCT). An event for this endpoint is death without evidence of disease progression or recurrence. Disease progression or recurrence will be considered competing events.
Grade 3+ Toxicities | Up to 2 years post transplant
  Adverse events and toxicities will be summarized using the NCI CTCAE v5.0. The person-year rates of Grade 3+ toxicity, grade 2-3 infections will be calculated with 95% CI.
Disease-Free Survival (DFS) | At 1 year
  Disease-free survival is the time from date of transplant to death or relapse/progression, whichever comes first. The event for this endpoint is relapse/progression or death.
  Participants alive and disease free will be censored at last available disease assessment.
Overall Survival (OS) | At 1 year and 2 years
  Overall survival is defined as the time interval between date of transplant and death from any cause. The event for this endpoint is death from any cause. Surviving participants will be censored at last follow-up.
Hematologic Recovery (Platelet Counts) | Up to 2 years post transplant
  Platelet recovery is defined by two different metrics: the first day of a sustained platelet count greater than or equal to 20,000/mm3 or greater than or equal to 50,000/mm3 with no platelet transfusions in the preceding seven days. The first day of sustained platelet count above these thresholds will be designated the day of platelet engraftment. The competing event is death or subsequent transplant without platelet recovery. For patients who never drop their platelet count below 20,000/mm3 or 50,000/mm3, the date of platelet recovery will be Day +1 post HCT.

CONTACTS AND LOCATIONS:
Overall Officials: Hannah Choe, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu